CLINICAL TRIAL: NCT00094081
Title: Phase III Randomized Trial of Concomitant Radiation, Cisplatin, and Tirapazamine Versus Concomitant Radiation and Cisplatin in Patients With Advanced Head and Neck Cancer
Brief Title: Concomitant Radiation and Cisplatin With and Without Tirapazamine in Treatment of Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC4690; SR259075
Record Dates: First submitted 2004-10-11; First posted 2004-10-14 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Head and Neck Neoplasms
Keywords: squamous cell carcinoma; oropharynx; oral cavity; larynx; hypopharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Laryngeal Diseases | interventions — Tirapazamine; Cisplatin; Radiotherapy

INTERVENTIONS:
Drug: tirapazamine (SR259075)
Drug: cisplatin
Procedure: Radiation Therapy

SUMMARY:
The trial will compare the efficacy and safety of concomitant chemoradiation with tirapazamine, cisplatin and radiation versus cisplatin and radiation.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx.
* Stage III or IV disease (excluding T1N1, and T2N1).
* ECOG performance status less than or equal to 2.
* Absolute neutrophil count at least 1.5 X 10^9/L, platelet count at least 100 X 10^9/L, and hemoglobin > 9g/dL.
* Serum bilirubin < 1.25 times ULN and AST/ALT < 2.5 times ULN.
* Calculated creatinine clearance (Cockcroft-Gault) > 55 mL/min.

Exclusion Criteria:

* Metastatic Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 861 (Actual)
Dates: Start 2002-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Overall survival.

SECONDARY OUTCOMES:
Time to locoregional failure.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (10):
- United States (10):
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Stanford University Medical Center, Palo Alto, California
  - H-Lee Moffitt Cancer Center and Research, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Harper Hospital, Detroit, Michigan
  - VA New Jersey Health Care Medical Center, East Orange, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - Eastern Virginia Medical School, Norfolk, Virginia

REFERENCES:
- [Derived] Ringash J, Fisher R, Peters L, Trotti A, O'Sullivan B, Corry J, Kenny L, Nuyts S, Wratten C, Rischin D. Effect of p16 Status on the Quality-of-Life Experience During Chemoradiation for Locally Advanced Oropharyngeal Cancer: A Substudy of Randomized Trial Trans-Tasman Radiation Oncology Group (TROG) 02.02 (HeadSTART). Int J Radiat Oncol Biol Phys. 2017 Mar 15;97(4):678-686. doi: 10.1016/j.ijrobp.2016.03.017. Epub 2016 Mar 23. PMID 27209505